CLINICAL TRIAL: NCT04588324
Title: Phase I/II Study Evaluating Safety and Clinical Efficacy of SHR2150 (TLR7 Agonist) in Combination With Chemotherapy Plus PD-1 or CD47 Antibody in Subjects With Unresectable/ Metastatic Solid Tumors
Brief Title: Study of SHR2150 (TLR7 Agonist) in Combination With Chemotherapy Plus PD-1 or CD47 Antibody in Subjects With Unresectable/ Metastatic Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Han weidong, Principal Investigator, Chinese PLA General Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-059
Record Dates: First submitted 2020-09-30; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Solid Tumor
Keywords: unresectable; metastatic; TLR7 agonist; anti-PD-1 antibody; anti-CD47 antibody; chemotherapy
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase 1 Dose-Escalation (Experimental): With a standard 3+3 dose escalation design, the enrollment will proceed until the MTD has been defined or the highest dose level has been reached.
  Interventions: Drug: SHR2150; Drug: Anti-Cancer Agent
- Phase 2 Dose-Expansion (Experimental): SHR2150 RP2D will be combined with chemotherapy plus PD-1 or CD47 antibody in 3-week treatment cycles.
  Interventions: Drug: Anti-Cancer Agent; Drug: SHR2150

INTERVENTIONS:
Drug: SHR2150 — Patients will receive escalating doses of SHR-2150 (starting dose 2 mg) in 3-week treatment cycles.
  Arms: Phase 1 Dose-Escalation
Drug: Anti-Cancer Agent — The previously resistant first-line cytotoxic regimens, anti-PD-1 antibody and/or anti-CD47 antibody will be administered intravenously Q3W.
Drug: SHR2150 — Patients will receive SHR-2150 at RP2D in 3-week treatment cycles.
  Arms: Phase 2 Dose-Expansion

SUMMARY:
This phase I/II trial aims to evaluate safety and efficacy of SHR2150 in combination with chemotherapy plus PD-1 or CD47 antibody in subjects with unresectable/ metastatic solid tumors. Patients will receive the combined regimen in 3-week treatment cycles. During the Phase 1 dose escalation portion of the trial, three oral doses of SHR2150 will be combined with intravenous administration of chemotherapy and PD-1 or CD47 antibody. In the Phase 2 dose expansion portion, patients will be treated with the Recommended Phase 2 Dose (RP2D) of SHR2150 in combination with chemotherapy plus PD-1 or CD47 antibody.

DETAILED DESCRIPTION:
Identification of T cell inhibitory signals, including PD-1/L1, has prompted the development of a new class of cancer immunotherapy that could restore an adequate immunosurveillance against the neoplasm and enhance T-cell-mediated anticancer immune responses. However, elimination of cancer by T cells is only one step in the cancer-immunity cycle, which enable providing several therapeutic targets and tailoring of combinations of immune therapies. SHR2150 is a small molecule agonist of toll-like receptors (TLRs) 7 designed to activate antigen-presenting cells and functions as mucosal immunoadjuvants in pre-clinical studies. This study is a first-in-man, Phase I/II, dose escalation/expansion study of a combined regimen of SHR2150 in combination with chemotherapy plus PD-1 or CD47 antibody in subjects with unresectable/ metastatic solid tumors. This study is designed to assess the safety, tolerability, RP2D and clinical efficacy of this regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have histologically proven unresectable/ metastatic solid tumors.
2. ≥ 18 years old.
3. Life expectancy of at least 6 months.
4. Eastern Cooperative Oncology Group performance status 0-3.
5. Subjects must have at least one measurable lesion ≥ 1 cm as defined by response criteria.
6. Subjects must have received at least two frontlines therapies, except for patients initially diagnosed with local advanced or metastatic pancreatic cancer or cholangiocarcinoma.
7. Subjects must be off prior therapy for at least 4 weeks prior to Day 1. Subjects with autologous hematopoietic stem-cell transplantation are eligible which must be more than 3 months. Subjects with Anti-PD-1 antibody are eligible which must be resistance.
8. Adequate organ function.
9. Female participants of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of study drug.
10. Male participants of childbearing potential must agree to use an adequate method of contraception, starting with the first dose of study drug through 120 days after the last dose of study drug.

Exclusion Criteria:

1. Subjects with any autoimmune disease or history of syndrome that requires corticosteroids or immunosuppressive medications.
2. Serious uncontrolled medical disorders or active infections, pulmonary infection especially.
3. Prior organ allograft.
4. Women who are pregnant or breastfeeding.
5. Women with a positive pregnancy test on enrollment or prior to investigational product administration.
6. Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-10-10 (Estimated); Primary Completion 2021-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Safety of the combined regimen of SHR2150, chemotherapy, PD-1 or CD47 antibody | 60 days after last dose
  Incidence, nature, and severity of adverse events graded according to the NCI CTCAE v5.0. AEs were considered to be treatment-related if they had started or worsened within the interval from first study drug administration until the follow-up visit.
Identify a RP2D of SHR2150 when given in combined regimen | 30 days
  The Recommended Phase 2 Dose (RP2D) of SHR2150 in the combined regimen will be identified at Phase 1 dose escalation period, and will be used in the phase 2 dose expansion period.
Object response rate (ORR) | 24 month
  ORR is defined as the proportion of subjects who achieved a partial response (PR) or complete response (CR) according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.

SECONDARY OUTCOMES:
Disease control rate (DCR) | 24 months
  DCR is defined as the proportion of subjects who achieved a stable disease (SD), partial response (PR) or complete response (CR) according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Progression-free survival (PFS) | 24 months
  PFS was measured from study entry to the first documentation of disease progression or death. Disease progression was determined per the RECIST V1.1.
Duration of Response (DOR) | 24 months
  DOR is defined as the time from the date of first documented response that is subsequently confirmed until date of documented progression or death in the absence of disease progression, the end of response should coincide with the date of progression or death from any cause used for the PFS endpoint. If the disease does not progress after a response, their duration of response will use the PFS censoring time.
Overall survival (OS) | 24 months
  OS was measured from the study entry to the date of death.
Time to Response (TTR) | 6 months
  TTR is defined as the period from the date of first dose to the date of the first evaluated response of CR or PR. If the response is not confirmed, it will not be included.

OTHER OUTCOMES:
Number of participants with laboratory test abnormalities | Approximately 6 months
  The bead-based immunoassay of serum cytokines and chemokines, such as IFN-α/β/γ, IL-6 and so on, will be performed on day 1 and 3 of each cycle, and the abnormality will be determined by the investigator.
Number of participants with pathological immunology marker change | Approximately 6 months
  Tumor tissues will be collected by biopsy at baseline and specified time points for all subjects. Tumor samples were analyzed by immunohistochemical pathological analysis and multiplex immunostaining.

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Han, Principal Investigator — Biotherapeutic Department of Chinese PLA General Hospital
Locations (1):
- Biotherapeutic Department of Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided